CLINICAL TRIAL: NCT03007628
Title: Magnetic Seizure Therapy Versus Electroconvulsive Therapy for Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14411961400
Record Dates: First submitted 2016-12-20; First posted 2017-01-02 (Estimated); Last update posted 2022-06-27 (Actual); Status verified 2022-05

CONDITIONS: Schizophrenia
Keywords: magnetic seizure therapy; electroconvulsive therapy; controlled trial
MeSH Terms: conditions — Schizophrenia | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- magnetic seizure therapy (Experimental): 10 treatment sessions of MST, three times per week in the first two weeks, two times per in the following two weeks.
  Interventions: Device: Magpro X100; Other: Treatment as usual (TAU)
- electroconvulsive therapy (Active Comparator): 10 treatment sessions of modified-ECT, three times per week in the first two weeks, two times per in the following two weeks.
  Interventions: Device: ThymatronSystem Ⅳ Electroconvulsive System; Other: Treatment as usual (TAU)

INTERVENTIONS:
Device: Magpro X100 — In addition to treatment as usual (TAU), participants are supposed to receive ten sessions of MST in four weeks, with three sessions per week in the first two weeks and two sessions per week in the following two weeks.
  Other Names: magnetic seizure therapy
  Arms: magnetic seizure therapy
Device: ThymatronSystem Ⅳ Electroconvulsive System — In addition to treatment as usual (TAU), participants are supposed to receive ten sessions of modified ECT in four weeks, with three sessions per week in the first two weeks and two sessions per week in the following two weeks.
  Other Names: electroconvulsive therapy
  Arms: electroconvulsive therapy
Other: Treatment as usual (TAU) — Participants will engage in their intpatient treatment program as-usual.

SUMMARY:
This trial attempts to evaluate the treatment efficacy of magnetic seizure therapy (MST) and its safety among schizophrenia patients. Half of the participants will be randomized to MST group, while the other half will be randomized to receive electroconvulsive therapy (ECT).

DETAILED DESCRIPTION:
Magnetic seizure therapy (MST) is likely to be an alternative options to electroconvulsive therapy (ECT).

Widespread stimulation of cortical and subcortical regions is inevitable for ECT since the substantial impedance of the scalp and skull shuts most of the electrical stimulus away from the brain. Nevertheless, magnetic pulses are capable to focus the stimulus to a specific area of the brain because they can pass the scalp and skull without resistance. In Addition, electric current will penetrate into deeper structures, while magnetic stimulus are only capable to reach a depth of a few centimeters. As a consequence, MST are able to generate focus stimuli on superficial regions of the cortex while ECT can't, which may give MST the capability to produce comparable therapeutic benefits with the absence of apparent cognitive side effects.

However, MST and ECT may both works via alterations of cortical inhibition and default mode network.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-5 diagnosis of schizophrenia;
2. convulsive therapy clinically indicated, such as severe psychomotor excitement or retardation, attempts of suicide, being highly aggressive, pharmacotherapy intolerance, and ineffectiveness of antipsychotics;
3. the positive and negative syndrome scale (PANSS)[20] score ≥ 60;
4. informed consent in written form.

Exclusion Criteria:

1. diagnosis of other mental disorders;
2. severe physical diseases, such as stroke, heart failure, liver failure, neoplasm, and immune deficiency;
3. present with a laboratory abnormality that could impact on efficacy of treatments or safety of participants;
4. failure to respond to an adequate trial of ECT lifetime;
5. are pregnant or intend to get pregnant during the study;
6. other conditions that investigators consider to be inappropriate to participate in this trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Changes in the Positive and Negative Syndrome Scale (PANSS) | At baseline and 4-week follow-up
changes in brain structure | At baseline, the 1 day after the first treatment, and at 4-week follow-up
  measured by Magnetic Resonance Imaging (MRI)

SECONDARY OUTCOMES:
Changes in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | At baseline and 4-week follow-up
Changes in Clinical Global Impressions (CGI) | At baseline and 4-week follow-up
Changes in motor threshold (MT) | At baseline and the day after the first treatment
  using single-pulse Transcranial Magnetic Stimulation (sTMS)
Changes in brain gamma-aminobutyric acid （GABA）levels | At baseline, between the first treatment and the second treatment, and at 4-week follow-up
  measured by Magnetic Resonance Spectroscopy (MRS)
Changes in resting state network (RSN) | At baseline, the day after the first treatment, and at 4-week follow-up
  measured by Magnetic Resonance Imaging (MRI)
Changes in auditory evoked potential (AEP) | At baseline and the day after the first treatment
  measured by electroencephalogram (EEG)
Changes in novel P300 potential | At baseline and the day after the first treatment
  measure by electroencephalogram (EEG)

CONTACTS AND LOCATIONS:
Overall Officials: Jijun Wang, PHD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD data